CLINICAL TRIAL: NCT05171192
Title: Feasibility Study of a Culturally Adapted Manual Assisted Brief Psychological Intervention (CMAP) Plus Learning Through Play (LTP) for Refugee Mothers with History of Self-harm in Pakistan
Brief Title: Culturally Adapted CMAP Plus LTP for Refugee Mothers with History of Self-harm in Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Collaborators: University of Manchester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SAHAR M-CMAP Plus LTP-002
Record Dates: First submitted 2021-12-11; First posted 2021-12-28 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Self-harm; Child Development
Keywords: Self-harm, Child development, Refugee mothers, CMAP, Learning through Play, LTP, Pakistan
MeSH Terms: conditions — Self-Injurious Behavior | interventions — Long-Term Potentiation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CMAP Plus LTP added to TAU (Experimental): C-MAP is a manual assisted intervention based on the principles of CBT which is focused on evaluation of the self-harm attempt, crisis skills, problem solving and basic cognitive techniques to manage emotions, negative thinking, and relapse prevention strategies. As family conflicts are a common issue with this group one session is focused on the use of culturally sensitive training in assertiveness and conflict management. The LTP is a community-based parenting intervention designed to deal with early child development. The central feature of the LTP intervention is a pictorial calendar devised for parents which depicts eight successive stages of child development from birth to 3 years along with illustrations of parent-child play and other activities that promote parental involvement, learning, and attachment.
  This will be added to Treatment as Usual
  Interventions: Behavioral: CMAP Plus LTP
- TAU alone (No Intervention): TAU alone will include routine follow up by Community Health Workers (CHWs) in Pakistan. Their work includes assisting with all aspects of maternal, new-born and childcare. Participants in treatment as usual arm will receive routine care.

INTERVENTIONS:
Behavioral: CMAP Plus LTP — The LTP Plus CMAP intervention will be delivered for a period of 12 weeks, including 8 weekly sessions and 2 sessions fortnightly. First 6 sessions will be for a duration of 60-90 minutes and remaining 4 sessions will take approximately 50-60 minutes. All sessions will be delivered by female therapists trained in CMAP and LTP intervention.
  Arms: CMAP Plus LTP added to TAU

SUMMARY:
Objectives:

* To asses the feasibility and acceptability of a culturally adapted manual assisted brief psychological intervention (CMAP) plus Learning through Play (LTP) for refugee mothers with history of self-harm having children 0-33 months. (Integrated intervention called CMAP Plus)
* To assess if CMAP Plus will reduce the repetition of self-harm in refugee mothers having children aged between 0-33 months.
* To determine if the intervention improves infant development and maternal attachment.
* To explore participants experiences with the intervention.

Study design and setting:

This will be a feasibility cluster randomized control trial (cRCT) of culturally adapted CMAP Plus LTP intervention with refugee mothers from Quetta and Peshawar, Pakistan.

Sample size:

We aim to recruit a sample of 80 refugee mothers in the study.

DETAILED DESCRIPTION:
Mental health of refugees particularly mothers living in camps or in conflict areas is one of the most important issues needing special attention and intervention. Culturally adapted Manual Assisted brief Psychological intervention (CMAP) utilizes problem solving components within a brief intervention that can be widely utilized in clinical practice in reducing repetition of self-harm in people who had recently self-harmed. Similarly, LTP programme promotes child health by supporting attuned interaction between mother and child, increasing maternal awareness of the physical and emotional needs of young children, and encouraging nurture and attachment. The CMAP plus LTP intervention may contribute significantly to the evidence base of addressing mental health of refugee mothers. This study aims to evaluate whether CMAP Plus LTP is feasible, acceptable for this population and helpful to reduce the repetition of self-harm and improve child development among refugee mothers with a history of self-harm. Eligible consented participants will complete the baseline assessments using structured questionnaires. Unit of randomization will be the Union Council. Uniion councils have been slected by the research team through consultations with community advisory committees from both sites. Selected UCs will be randomized into two study arms: 1) C-MAP plus LTP added to treatment as usual and 2) Treatment as usual (TAU) alone. Participants in intervention arm will receive 10 individual sessions of CMAP plus LTP intervention for a period of 12 weeks. All sessions will be delivered by female therapists trained in CMAP Plus. Participants in TAU alone group will receive routine care that includes routine follow up by Community Health Workers (CHWs) in Pakistan. Assessments will be carried out at baseline, and completion of the intervention at 12th week (after intervention). All assessments will be rater-blind (done by independent RAs (female), not involved in delivering the intervention sessions). After post-assessments, a purposefully selected subset (stratified by age) of participants will be invited for qualitative interviews (n = up to 15 interviews) to explore their experiences and satisfaction with the intervention. On average, interviews will last for 60-90 minutes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above refugee mothers with children aged between 0-33 months.
* History of self-harm.
* Resident in the study site.
* Capacity to provide informed consent.
* Available for the duration of the study.

Exclusion Criteria:

* Unable to provide consent due to severe mental or physical illness.
* Unlikely to be available for the entire duration of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Refugee mothers with children aged between 0-33 months
Enrollment: 80 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Feasibility measure | From baseline to 12th week (at the end of intervention)
  The feasibility will be determined by collating data on recruitment and retention rates. The success criterion of feasibility will be to recruit > 50% of eligible participants.
Acceptability measure | From baseline to 12th week (at the end of intervention)
  The intervention acceptability will be assessed using data on attendance. Criterion for acceptability is a mean attendance rate of >70% of at least 7 sessions.

SECONDARY OUTCOMES:
Suicide Attempt Self-Injury Interview | From baseline to 12th week
  Repetition rate of self-harm at 3 months after randomisation as measured by adapted Suicide Attempt Self-Injury Interview. The questionnaire records self-harm events by severity and chronological order.
Beck Scale for Suicide Ideation | Change in problem scores from baseline to 12th week
  This is a 19-item instrument for detecting and measuring the current intensity of the patients' specific attitudes, behaviours, and specificity of a patient's thoughts to kill him/herself during the past week.
Beck Depression Inventory | Change in problem scores from baseline to 12th week
  This is a 21 items scale measuring symptoms of depression. Higher scores on the scale indicate greater severity of depression.
Beck Hopelessness Scale | Change in problem scores from baseline to 12th week
  This instrument is designed to measure three aspects of hopelessness, feelings about the future, loss of motivation and expectations.
Generalized Anxiety Disorder | Change in problem scores from baseline to 12th week
  This is a 7-item scale used to screen for and measure severity of Generalized Anxiety Disorder.
Assessment of the growth and development of children | Change from baseline to 12th week
  Anthropometric measures of child growth will be collected through measuring children's height, weight and head circumference
Ages and Stages Questionnaire and ASQ Socio-emotional Scales | Change from baseline to 12th week
  Ages and Stages Questionnaire and ASQ Socio-emotional scales will be used to measure child development. Parents will report on their child's communication, gross motor, fine motor, problem solving and personal-social development at different time points.
Coping resource inventory | Change from baseline to 12th week
  Coping resource inventory will assess the coping resources to manage stress available to an individual.
Problem Solving Inventory | Change in problem scores from baseline to 12th week
  The Problem-Solving Inventory assesses an individual's awareness and evaluation of his or her problem-solving abilities or styles. The problem-solving Inventory is a self-report measure, and thus assesses perceptions of problem solving as opposed to actual problem-solving skills.
Infant Development Questionnaire | Change from baseline to 12th week
  Infant Development Questionnaire is a 20-item questionnaire of paternal knowledge and expectations for child development in the first three years.
Parenting Stress Index - Short Form | Change from baseline to 12th week
  Parents rated 36 item scale on five-point scale (1-5). The scale consists of three subscales: (1) Parenting Distress, (2) Difficult Child Characteristics, and (3) Dysfunctional Parent-Child Interaction.
Multidimensional Scale of Perceived Social Support | Change from baseline to 12th week
  This brief scale will assess perceived social support.
Euro-Qol-5 Dimensions scale | Change in problem scores from baseline to 12th week
  Health-related quality of life will be measured using the Euro-Qol-5 Dimensions scale. This is a standardized instrument that measures five health dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each scored from 1 to 3 indicating "no problem" to "severe problems".
Client Service Receipt Inventory | Change from baseline to 12th week
  This inventory will collect information about the use of other health services (including the informal sector faith healers/Imams) using CSRI based on our previous work in Pakistan
Client Satisfaction Questionnaire | Change from baseline to 12th week
  The participants will rate their satisfaction with treatment using the Client Satisfaction Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Nusrat Husain, Principal Investigator — University of Manchester; Nasim Chahudhry, Principal Investigator — Pakistan Institute of Living and Learning
Locations (2):
- Pakistan (2):
  - Community Settings, Quetta, Balochistan
  - Community settings, Peshawar, KPK

IPD SHARING:
Plan to Share IPD: No